CLINICAL TRIAL: NCT00951184
Title: Efficiency of Screening for Depression in Cancer Patients Receiving Radiotherapy
Brief Title: Depression Screening in Patients Undergoing Radiation Therapy For Cancer
Status: Completed | Type: Observational
Sponsor: Radiation Therapy Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH); NRG Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: RTOG 0841; CDR0000643316
Record Dates: First submitted 2009-08-01; First posted 2009-08-04 (Estimated); Last update posted 2015-03-18 (Estimated); Status verified 2015-03

CONDITIONS: Depression; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: depression; unspecified adult solid tumor, protocol specific
MeSH Terms: conditions — Depression | interventions — Psychiatric Rehabilitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: telephone-based intervention
Other: screening questionnaire administration
Other: study of socioeconomic and demographic variables
Procedure: assessment of therapy complications
Procedure: psychosocial assessment and care

SUMMARY:
RATIONALE: Gathering information about depression in patients with cancer may help doctors learn more about the disease and plan the best treatment.

PURPOSE: This clinical trial is studying depression screening in patients undergoing radiation therapy for cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Assess the feasibility of a screening procedure for major depression in cancer patients undergoing definitive or palliative radiotherapy.

Secondary

* Establish the rates of major depression identified through diagnostic telephone interviews.
* Estimate the false negative rate (1-sensitivity) and false positive rate (1-specificity) of the 9-item Patient Health Questionnaire (PHQ-9) and the 25-item Hopkins Symptom Checklist (HSCL-25).
* Compare the false negative rate of 2 items addressing mood disturbance on the PHQ-9 relative to all 9-items on the PHQ-9 and to the HSCL-25.
* Examine the sensitivity to changes in depression severity of the PHQ-9, the HSCL-25, and the Structured Clinical Interview for DSM-IV (SCID) .
* Correlate both depressive symptoms and major depression in terms of sociodemographic and clinical variables.
* Establish the nature and adequacy of existing care, patient preferences, treatment availability, and barriers to depression treatment utilization for patients identified with major depression using the Assessment of Mental Health Services and Barriers to Care.
* Assess rates of continued elevations of depressive symptoms, seeking and receipt of care, and barriers to care at follow-up in these patients.
* Examine the differences in study objectives based on institution characteristics with regard to existing psychosocial services that are provided on-site and integrated in cancer care.

OUTLINE: This is a multicenter study.

* Depression screening: Patients complete screening depression questionnaires, including the Hopkins Symptom Checklist (HSCL-25) and the 9-item Patient Health Questionnaire (PHQ-9) that includes a 2-item PHQ, and a Health Status Questionnaire at baseline.
* Diagnostic telephone interview: Within 2 weeks, patients who screen positive for depression and select patients who screen negative for depression undergo a diagnostic telephone interview that includes modules of the Structured Clinical Interview for Diagnosis-DSM-IV (SCID) related to major depression, bipolar disorder, adjustment disorders, and queries concerning past and current mental health treatment and barriers to treatment. The Assessment of Mental Health Services and Barriers of Care questionnaire is also administered by the clinical interviewer. Clinical interviewers provide patients who are found to be depressed with a list of community resources, and offer assistance in obtaining treatment, if needed. Patients are also encouraged to discuss these options with their oncology health care team.
* Follow-up interview: At 3 months, patients who receive a research diagnosis of major depression, dysthymia, bipolar disorder, or cancer-related adjustment disorder in the initial SCID-DSM-IV undergo another diagnostic telephone interview and are reassessed for the initiation and continuation of treatment, current depressive symptoms, and receipt of cancer care. The HSCL-25, PHQ-9, and Assessment of Mental Health Services and Barriers of Care questionnaires and the SCID-DSM-IV are also administered by the clinical interviewer. Treatment options and referrals are discussed with patients who remain depressed and are not in treatment.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of any tumor type

  * Scheduled to begin radiotherapy within 2 weeks
  * Stage I-IV cancer (where applicable) allowed
* Pre-existing diagnosis of depression allowed

PATIENT CHARACTERISTICS:

* Zubrod performance status 0-1
* Able to speak and read English sufficiently to complete screening instruments
* Must have existing land-line or cellular telephone service
* Not considered suicidal, psychotic, or otherwise unfit for study participation by cancer center staff clinical judgment
* No concurrent medical or psychiatric condition that, in the opinion of the investigator, would potentially pose a risk to the patient as a result of participation in this trial
* Not mentally incompetent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Prior or concurrent combination therapy with surgery, chemotherapy, hormone therapy, or immunotherapy allowed
* No concurrent psychotropic medication, psychotherapy, or pharmacotherapy for depression at screening
* Not receiving hospice care

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult (at least age 21) cancer patients who are undergoing radiation therapy for their first diagnosis of cancer with no mental incompetence which would preclude completion of questionnaires, who is not considered suicidal or psychotic or otherwise unfit for study participation. Patient must provide study-specific consent prior to screening.
Sampling Method: Non-Probability Sample
Enrollment: 463 (Actual)
Dates: Start 2009-05; Primary Completion 2011-10 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Feasibility of a screening procedure for major depression | Within 1 week of registration

SECONDARY OUTCOMES:
Rates of major depression as identified in diagnostic telephone interviews | Within 4 weeks of registration
False negative rate and false positive rate of the 9-item Patient Health Questionnaire (PHQ-9) and the 25-item Hopkins Symptom Checklist (HSCL-25) | Within 4 weeks of registration
False negative rate of 2 items addressing mood disturbance on the PHQ-9 relative to all 9-items on the PHQ-9 and to the HSCL-25 | Within 4 weeks of registration
Sensitivity to changes in depression severity of the PHQ-9, the HSCL-25, and the Structured Clinical Interview for DSM-IV (SCID) | Within 4 weeks of registration
Sociodemographic and clinical correlates with depressive symptoms and major depression | Within 4 weeks of registration
Patient preferences, existing care, treatment availability, and barriers to its utilization determined at the diagnostic interview | Within 4 weeks of registration
Symptoms, seeking and receipt of care, and barriers to care at 3-month follow-up | Within 4 weeks of registration
Differences in study endpoints based on institution characteristics with regard to existing psychosocial services that are provided on-site and integrated in cancer care | Within 1 week of registration

CONTACTS AND LOCATIONS:
Overall Officials: Lynne Wagner, MD, Principal Investigator — Robert H. Lurie Cancer Center
Locations (16):
- United States (16):
  - Saint Anthony's Hospital at Saint Anthony's Health Center, Alton, Illinois
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - CCOP - Grand Rapids, Grand Rapids, Michigan
  - St. John's Regional Health Center, Springfield, Missouri
  - Hulston Cancer Center at Cox Medical Center South, Springfield, Missouri
  - David C. Pratt Cancer Center at St. John's Mercy, St Louis, Missouri
  - CCOP - North Shore University Hospital, Manhasset, New York
  - Long Island Jewish Medical Center, New Hyde Park, New York
  - Mission Hospitals - Memorial Campus, Asheville, North Carolina
  - Pardee Memorial Hospital, Hendersonville, North Carolina
  - FirstHealth Moore Regional Community Hospital Comprehensive Cancer Center, Pinehurst, North Carolina
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Cancer Center of Paoli Memorial Hospital, Paoli, Pennsylvania
  - Lankenau Cancer Center at Lankenau Hospital, Wynnewood, Pennsylvania
  - St. Mary's Hospital Medical Center - Green Bay, Green Bay, Wisconsin
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin